CLINICAL TRIAL: NCT02014688
Title: Multi-center Study for Normal Database of Optic Nerve Head, Retinal Nerve Fiber Layer, and Macula Parameters With the Heidelberg Spectralis OCT, Study 3
Brief Title: Optical Coherence Tomography (OCT) Normative Data Collection Study
Acronym: S-2013-3
Status: Completed | Type: Observational
Sponsor: Heidelberg Engineering GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: S-2013-3 NORM-us
Record Dates: First submitted 2013-12-11; First posted 2013-12-18 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Healthy
Keywords: Normal subjects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- American Indian or Alaskan Native Descent
- Black or African American Descent
- Asian Descent
- Hispanic Descent

SUMMARY:
This study is being initiated to create a normal database including measures of optic nerve head (ONH), peripapillary retinal nerve fiber layer (RNFL), and macula using the Heidelberg Spectralis OCT device.

DETAILED DESCRIPTION:
This multi-center, prospective, observational (non-interventional) study is the third in a series to measure structural parameters of the optic nerve head, the peripapillary retinal nerve fiber layer, and the macula using the Heidelberg Spectralis OCT device. This study is conducted in normal volunteers of various non-Caucasian ethnic group, and data will be combined with Caucasian subjects to be representative of the US population: (1) Hispanic Descent, (2) Black or African American Descent, (3) Asian Descent, (4) American Indian or Alaskan Native Descent. This study will complement the previous study S-2012-1 NORM-cc, in which normal data from Caucasian individuals were collected.

The main goal of the study is to provide the range of these structural parameters in normal eyes. The study will include at least 87 (enrollment target: 135) normal volunteers; each study site will recruit at least 29 (target: 45) subjects with an age range of 18 to 90 years and an approximately equal number of females and males. All subjects will undergo Spectralis OCT imaging, biometric and ophthalmoscopic examination, disc photography and visual field testing in one single visit. All examinations performed on the subjects are non-significant risk procedures because the medical devices are cleared for marketing in Europe and in the U.S. Total study duration including IRB approval is anticipated to not exceed 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Subject is not an employee of the eye clinic.
* Age ≥18 to 90.
* Able and willing to undergo the test procedures, give consent, and to follow instructions.
* Healthy eye without prior intraocular surgery (except cataract surgery) and without clinically significant vitreal, retinal or choroidal diseases, clinically significant diabetic retinopathy (subject may have diabetes), or disease of the optic nerve. Small Drusen are acceptable in older subjects.
* Hispanic Descent, Black or African American Descent, Asian Descent, American Indian or Alaskan Native Descent
* Negative history of glaucoma.
* Intraocular pressure ≤21mmHg.
* Best corrected visual acuity ≥0.5.
* Refraction between +6 and -6 diopters and astigmatism ≤ 2 diopters.
* Normal visual field with Glaucoma Hemifield Test and Mean Deviation within normal limits, or not abnormal visual field by judgment of the ophthalmologist.
* Clinically normal appearance of the optic disc, with normal appearing neuroretinal rim with respect to color and shape. The optic disc is examined ophthalmoscopically and by evaluation of stereo photographs.
* When both eyes are eligible, both eyes enter the study.

Exclusion Criteria:

* Unreliable visual field. The reliability indices should be used as guide as well as the perimetrist's notes.
* Unusable disc stereo photos.
* Inability to undergo the tests.
* Insufficient quality of Spectralis OCT images (this is not determined until after Spectralis OCT examination, and is an unusual circumstance). Minimum requirements are:

  * Retina completely included in image frame,
  * Quality Score ≥ 20 in the stored ART mean images, and
  * For ONH-R scan: Center position error ≤ 100 μm.
* Note: Inability of a subject to perform one of the two scan patterns or insufficient image quality in one scan pattern does not exclude the subject or eye from the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recruitment will be from persons who respond to recruitment initiatives at the individual centers or have signed a release saying that they are willing to be approached for participation in research.
  At least 87 subjects (enrollment target: 135 subjects) will be selected from qualifying normal volunteers. Age range will be from ≥18 to 90 years. The age of the subjects will be defined by their month of birth versus the month of giving consent to participate in this study. A subject who is 40 years and 11 months old will be counted as being in the age group "31 to 40 years". Each site will attempt to recruit subjects in about equal numbers in each age group. The distribution in the age groups should be fairly equal among subjects in each ethnic group alone.
Sampling Method: Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2013-12; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Normative Data for optic nerve head, the peripapillary retinal nerve fiber layer, and the macula. | 12 months
  This normal database will be used to determine if an unknown subject has measurement values "within normal limits" or "outside normal limits." It is planned to classify an eye "within normal limits" if the measurement value is greater than or equal to the 5th percentile of the normal distribution (or less than or equal to the 95th percentile), and as "outside normal limits" if the measurement value is smaller than the 1st percentile (or larger than 99th percentile) of the normal distribution. Thus, the sample size must be large enough to ensure that the 1st and the 5th percentiles of the distribution are distinct.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Liebman, MD, Principal Investigator — Manhattan Eye, Ear and Throat Hospital and New York University Medical Center
Locations (1):
- New York Eye and Ear Infirmary, New York, New York, United States